CLINICAL TRIAL: NCT05943925
Title: Dementias and Microbiota Composition: Is Possible to Revert the Dementia Symptoms Reverting the Microbiota Composition?
Acronym: DEM-BIOTA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Rovira i Virgili (Other)
Collaborators: Ministerio de Ciencia e Innovación, Spain (Other Government)
Responsible Party: Principal Investigator, Margarita Torrente, Dr., University Rovira i Virgili
Other Study IDs: PID2019-103888RB-I00
Record Dates: First submitted 2023-04-26; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-06

CONDITIONS: Dementia Alzheimers; Dementia With Lewy Bodies; Parkinson Disease Dementia; Dementia Frontotemporal; Mild Cognitive Impairment
Keywords: cognitive status; functional status; neuropsychiatric status; microbiota
MeSH Terms: conditions — Alzheimer Disease; Lewy Body Disease; Pick Disease of the Brain; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — stool sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Healthy control group: The criteria for the recruitment will be:
  Inclusion criteria: more than 60 years. Exclusion criteria: Significant neurology disease diagnosed, infectious treatment with antibiotics in the previous 6 months prior to providing the stool sample, corticosteroid use, immunosuppressors or immunostimulants treatment, illnesses of the gastrointestinal (GI) tract, large doses of commercial probiotics consumed (greater than or equal to 108 colony forming units (cfu) per organisms per day).
  This control group were recruited from relatives of the patients enrolled or general population and interviewed at the hospital (relatives, University or their homes).
  Neuropsychological, functional and neuropsychiatric assessment and stool sample.
  Interventions: Other: No intervention
- Alzheimer Disease (AD): The criteria for the recruitment will be:
  Inclusion criteria: Alzheimer Disease (AD) diagnosed by the neurology service; more than 60 years.
  Exclusion criteria: Comorbidity with other significant neurology disease, infectious treatment with antibiotics in the previous 6 months prior to providing the stool sample, corticosteroid use, immunosuppressors or immunostimulants treatment, illnesses of the GI tract, large doses of commercial probiotics consumed (greater than or equal to 108 colony forming units (cfu) per organisms per day).
  Neuropsychological, functional and neuropsychiatric assessment and stool sample.
  Interventions: Other: No intervention
- Mild Cognitive Impairment (MCI)- amnesic: The criteria for the recruitment will be:
  Inclusion criteria: Mild Cognitive Impairment (MCI) amnesic, diagnosed by the neurology service; more than 60 years.
  Exclusion criteria: Comorbidity with other significant neurology disease, infectious treatment with antibiotics in the previous 6 months prior to providing the stool sample, corticosteroid use, immunosuppressors or immunostimulants treatment, illnesses of the gastrointestinal (GI) tract, large doses of commercial probiotics consumed (greater than or equal to 108 colony forming units (cfu) per organisms per day).
  Neuropsychological, functional and neuropsychiatric assessment and stool sample.
  Interventions: Other: No intervention
- Parkinson Disease Dementia (PDD): The criteria for the recruitment will be:
  Inclusion criteria: Parkinson Disease Dementia (PDD) diagnosed by the neurology service; more than 60 years.
  Exclusion criteria: Comorbidity with other significant neurology disease, infectious treatment with antibiotics in the previous 6 months prior to providing the stool sample, corticosteroid use, immunosuppressors or immunostimulants treatment, illnesses of the gastrointestinal (GI) tract, large doses of commercial probiotics consumed (greater than or equal to 108 colony forming units (cfu) per organisms per day).
  Neuropsychological, functional and neuropsychiatric assessment and stool sample.
  Interventions: Other: No intervention
- Lewy bodies dementia (LBD): The criteria for the recruitment will be:
  Inclusion criteria: Lewy Body Dementia (LBD) diagnosed by the neurology service; more than 60 years.
  Exclusion criteria: Comorbidity with other significant neurology disease, infectious treatment with antibiotics in the previous 6 months prior to providing the stool sample, corticosteroid use, immunosuppressors or immunostimulants treatment, illnesses of the gastrointestinal (GI) tract, large doses of commercial probiotics consumed (greater than or equal to 108 colony forming units (cfu) per organisms per day).
  Neuropsychological, functional and neuropsychiatric assessment and stool sample.
  Interventions: Other: No intervention
- Frontotemporal Dementia (FTD)-behavioral variant: The criteria for the recruitment will be:
  Inclusion criteria: Frontotemporal Dementia (FTD)-behavioral variant diagnosed by the neurology service; more than 60 years.
  Exclusion criteria: Comorbidity with other significant neurology disease, infectious treatment with antibiotics in the previous 6 months prior to providing the stool sample, corticosteroid use, immunosuppressors or immunostimulants treatment, illnesses of the gastrointestinal (GI) tract, large doses of commercial probiotics consumed (greater than or equal to 108 colony forming units (cfu) per organisms per day).
  Neuropsychological, functional and neuropsychiatric assessment and stool sample.
  Interventions: Other: No intervention
- Alzheimer disease (AD)-control: Inclusion criteria: Alzheimer Disease (AD) diagnosed by the neurology service; more than 65 years. Exclusion criteria: Comorbidity with other significant neurology disease, infectious treatment with antibiotics in the previous 6 months prior to providing the stool sample, corticosteroid use, immunosuppressors or immunostimulants treatment, illnesses of the gastrointestinal (GI) tract, large doses of commercial probiotics consumed (greater than or equal to 108 colony forming units (cfu) per organisms per day).
  Neuropsychological, functional and neuropsychiatric assessment and stool sample at basal, 12 weeks and 24 weeks.
  Interventions: Dietary Supplement: Probiotic supplement
- Alzheimer disease (AD)-probiotic: Inclusion criteria: Alzheimer Disease (AD) diagnosed by the neurology service; more than 65 years. Exclusion criteria: Comorbidity with other significant neurology disease, infectious treatment with antibiotics in the previous 6 months prior to providing the stool sample, corticosteroid use, immunosuppressors or immunostimulants treatment, illnesses of the gastrointestinal (GI) tract, large doses of commercial probiotics consumed (greater than or equal to 108 colony forming units (cfu) per organisms per day).
  Neuropsychological, functional and neuropsychiatric assessment and stool sample at basal, 12 weeks and 24 weeks.
  Interventions: Dietary Supplement: Probiotic supplement

INTERVENTIONS:
Other: No intervention — no intervention
  Groups: Alzheimer Disease (AD); Frontotemporal Dementia (FTD)-behavioral variant; Healthy control group; Lewy bodies dementia (LBD); Mild Cognitive Impairment (MCI)- amnesic; Parkinson Disease Dementia (PDD)
Dietary Supplement: Probiotic supplement — A total of 60 Alzheimer Disease (AD) patients will be recruited, 30 will ingest the probiotic mixture and 30 will ingest placebo (randomized assignment to the groups will be done). The experimental group will take the probiotic ingest daily: Lactobacillus acidophilus, Lactobacillus casei, Bifidobacterium bifidum, and Lactobacillus fermentum (2 × 109 colony forming units (CFU)/g of each). This mixture of bacteria has been showed to have positive results with 12 weeks treatment.
  Groups: Alzheimer disease (AD)-control; Alzheimer disease (AD)-probiotic

SUMMARY:
Dementia is the major cause of disability and dependency among older adults worldwide affecting memory, cognitive abilities and behavior, interfering with one's ability to perform daily lives activities. Although age is the strongest known risk factor for the onset of dementia, it is not a natural or inevitable consequence of aging. Dementia not only affects older people, since up to 9% of the cases appear before 65 years. The impact of dementia is highly important in financial terms also in human costs to countries, societies and individuals.

Dementia is an umbrella term for several diseases, being Alzheimer's disease (AD) the most common form, contributing to 60-70% of cases. Other major forms include Lewy bodies Dementias (LBDs) and frontotemporal dementia (FTD).

The role of the gastrointestinal microbiota in human brain development and function is an area of increasing interest and research. A large number of studies suggest that the gut microbiota can influence the brain, cognition and behavior of the patients, and also modulate brain plasticity, modifying brain chemistry via various mechanisms like neural, immune and endocrine Within these last two years some studies have showed differences in the microbiota of the AD patients from healthy controls. In this sense, increasing number of studies, most of them in animal models, support the notion that probiotics have significant benefit in maintaining homeostasis of the Central Nervous System. And recent studies try to replicate this finding in AD patients with controversial results.

The main objective of DEM-BIOTA project is to improve the knowledge of the relationship between microbiota and dementia. DEM-BIOTA will explore the microbiota differences between dementias: AD, LBDs, that includes: Parkinson disease dementia (PDD) and Lewy Body Dementia (LBD) and FTD-behavioral variant, also in Mild Cognitive Impairment (MCI) to study the progression; in our context (Mediterranean diet and lifestyle) and characterize them in relation to neurocognitive and neuropsychiatric symptoms as well as patient functionality (dependency level). Moreover, the capacity of a probiotic compound in reverting or improving neurocognitive and neuropsychiatric symptoms and patient functionality in a sample of AD patients will be also studied.

DETAILED DESCRIPTION:
Hypothesis: Currently any other study to our knowledge has studied the relationship between gut microbiota and dementia symptoms in our country. Although there are few recent studies that have explored relations between microbiota and dementia, they were conducted in Japan or USA. Taken into account the important factor of diet and lifestyle in microbiota composition and the differences between these countries (Japan and USA) and Mediterranean diet and lifestyle, it was the need of a relational study in our context. The hypothesis is that although it will be different microbiota between healthy and demented subjects, the microbiota composition of healthy subjects in Mediterranean context could significant differ from the above-mentioned studies.

In the few studies already conducted, the patients included were diagnosticated of AD or it were included patients from all type of dementias. Even though AD is the most common type of dementia, there are more types of dementias that should be considered differentially as the features are significantly different. Given the diversity through the symptoms across dementias, a characterization of the gut microbiota of different types of dementia will be described, specifically, AD, LBDs: LBD and PDD separately, and FTD-behavioral variant. Furthermore, MCI subjects will be also studied in order to explore the microbiota changes before the onset of dementia (taking into account the high percentage of MCI that progress to dementia). These studies could reveal a risk factor compositional microbiota to develop dementia. The hypothesis is that microbiota will differ through different dementias and could be related to the feature symptoms of each one, being MCI subjects between healthy and dementia patients, in terms of microbiota composition.

As pointed out in the introduction, preclinical research shows that probiotics may improve cognitive performances in animal models with impaired cognition. However, data about the effects of probiotics on cognitive performance or psychopathological symptoms in humans are scarce and controversial. This lack of agreement could due to the differences in the population studied (young adults, elderly, healthy and clinic population, neurologic and psychiatric patients), the measures (different mood scales and different cognitive assessments), the probiotic compositions and the duration of treatment (from 3 weeks to 12 weeks). Considering the lack of knowledge about the probiotics potential treating dementia symptoms, dementia AD patients will be treated with a probiotic compound (a probiotic mixture already successful in improving cognitive impairment in AD patients, but only assessed by a cognitive screening and with no analysis of microbiota). The study will be conducted in an elderly group affected from AD, with a broad type of neuropsychological, neuropsychiatric and functional measures, and microbiota characterization at 12 and 24 weeks of treatment. An improvement of dementia symptoms due to probiotic consumption is expected, not only neuropsychological but also at a neuropsychiatric and functional level and these changes will be related to the changes of microbiota composition.

General objective: The main objective of DEM-BIOTA is to confirm the relationship between microbiota and dementia in our model of diet and lifestyle, improving the knowledge of the relationship between microbiota and dementias. This means to explore the possible differences between dementias in relation to microbiota in our context (Mediterranean diet and style of life) and characterize them in relation to neurocognitive and neuropsychiatric symptoms as well as patient functionality (dependency level). Moreover, the capacity of a probiotic compound in reverting or improving neurocognitive and neuropsychiatric symptoms and patient functionality will be studied.

This objective will be achieved through a multidisciplinary study considering microbiota composition and deep study of the dementia symptoms taking into account the personal characteristics of each patient. The final issue is to draw a relational map about the microbiota composition and dementia symptoms and the identification of the microbiota strains that are a risk factor of produce a deficit in metabolites. The project proposes to finally study how can a probiotic mixture improve AD symptoms, and study in deep the microbiota composition changes along with the changes (or not) of dementia symptoms.

This main objective will be carried out by combining our previous knowledge, partly of the collaboration with European Union partners, with data provided by literature on international studies on human population.

The aim match with the activities addressed in 1st Challenge identified in the Spanish Strategy for R+D+I Targeted to Societal Challenges "Health, Geographical change and Well-being": 1.1.2. Understanding disease; 1.2.1. Development of effective prevention and detection programs and improvement of disease propensity assessment.

1.3. SPECIFIC OBJECTIVES

1. - Protocol revision and preparation. Revision of the all tests and scales, writing down all the protocols, alignment the study protocols with the hospitals' procedures, timetables, sample collection protocols, etc.
2. - Study the microbiota composition (from stool samples of the patients) of AD patients in our context (Mediterranean lifestyle).

   Describe the microbiota composition from AD patients in relation with their healthy controls.

   To what extent does it differ from their controls and from the AD patient's composition of other countries?
3. - Study microbiota composition differences (from stool samples of the patients) between some of the most known dementias: AD, PDD, LBD, FTD-behavioral variant

   Describe and compare microbiota composition between some of the most known dementias: AD, PDD, LBD, FTD-behavioral variant.

   Describe and compare microbiota composition between MCI patients and AD patients.

   Describe and compare microbiota composition between MCI patients and PDD, LBD, FTD-behavioral variant patients.

   Are there any relations between the microbiota composition of all experimental groups with neuropsychological, neuropsychiatric and functional characteristics present in these dementias and in these patients? All these relations could be modulated by life stressors and diet (adherence to Mediterranean diet)?
4. - Study the effects of a probiotic compound in AD patients. In relation to AD symptoms: neuropsychological, neuropsychiatric and functional In relation to microbiota composition (analyzed from the stool samples of the patients) Until what extend and how the microbiota composition explains the AD symptoms? Can this probiotic compound improve the symptoms and is in general a good treatment/complement to the nowadays treatment?
5. - Dissemination and formation. Dissemination of results at scientific (open access journals, congresses and other national and international meetings) and social level disclosure (newspapers, research group web, webs of the hospitals and Alzheimer association, conferences to general public, radio, television, etc.), as well as formation to patients, professionals and general public.

ELIGIBILITY:
Inclusion Criteria:

Study 1, microbiota composition study- AD, PD, LBD, FTD-behavioral variant or MCI-amnesic

* diagnosed by the neurology service (or healthy subjects, without any of these diagnostics).
* more than 60 years

Study 2-probiotic intervention,:

* AD diagnosed by the neurology service;
* more than 65 years.

Exclusion Criteria:

Study 1, microbiota study:

* Comorbidity with other significant neurology disease,
* Infectious treatment with antibiotics in the previous 6 months prior to providing the stool sample,
* corticosteroid use,
* immunosuppressors or immunostimulants treatment,
* illnesses of the Gastro Intestinal tract,
* large doses of commercial probiotics consumed (greater than or equal to 10 elevated to 8 colony forming unit per organisms per day).

Study 2-probiotic intervention:

* Comorbidity with other significant neurology disease,
* Infectious treatment with antibiotics in the previous 6 months prior to providing the stool sample,
* corticosteroid use,
* immunosuppressors or immunostimulants treatment,
* illnesses of the GI tract,
* large doses of commercial probiotics consumed (greater than or equal to 10 elevated to 8 cfu per organisms per day).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinic patients from hospitals and other diagnostic medical centers.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Shotgun sequencing metagenomics analysis (NextSeq2000) | Baseline for all the group subjects subjects in microbiota composition study. Baseline, change from baseline at 12 weeks and change from baseline at 24 weeks for Alzheimer Disease (AD) patients in the probiotic study.
  Gut microbiome was analysed using a shotgun metagenomic approach. DNA was extracted from samples using the DNA Preparation with Tagmentation kit, according to manufacturer protocols (Illumina, California, USA, catalog no. 20018705). Sequencing libraries concentration was determined by Qubit 4.0 fluorometer and Qubit dsDNA High Sensivity Assay Kit (Thermo Fisher Scientific, Massachusetts, USA). Sequencing libraries length was checked by Agilent TapeStation and Agilent High Sensitivity DNA kit (Agilent Technologies, California, USA). Sequencing libraries with concentration below 750 per Molar and length out of 400-600 bp range were discarded. Final sequencing libraries were mixed at 750 bp and sequenced using the NextSeq 2000 sequencing system (Illumina, California, USA) as 2x150-bp paired-end reads. Samples below 7,5 million reads were discarded. Shotgun metagenomic reads were profiled for microbial species relative abundances by mapping them to several databases with Kraken2.
Neuropsychology assessment: Mini Mental State Examination (MMSE) | Baseline for all the group subjects subjects in microbiota composition study. Baseline, change from baseline at 12 weeks and change from baseline at 24 weeks for AD patients in the probiotic study.
  Mini Mental State Examination (MMSE), screening test for cognitive deterioration.
  At Baseline for no intervention study, study 1.
  For the probiotic study, study 2, at baseline, change at 12 weeks and change at 24 weeks
Neuropsychology assessment: Global Deterioration Scale-Functional Assessment Staging (GDS-FAST) | Baseline for all the group subjects subjects in microbiota composition study. Baseline, change from baseline at 12 weeks and change from baseline at 24 weeks for AD patients in the probiotic study.
  Global Deterioration Scale-Functional Assessment Staging (GDS-FAST)
  At Baseline for no intervention study, study 1.
  For the probiotic study, study 2, at baseline, change from baseline at 12 weeks and change from baseline at 24 weeks.
Neuropsychology assessment: Clinical Dementia Rating (CDR) | Baseline for all the group subjects subjects in microbiota composition study. Baseline, change from baseline at 12 weeks and change from baseline at 24 weeks for AD patients in the probiotic study.
  Clinical Dementia Rating (CDR) score.
  At Baseline for no intervention study, study 1.
  For the probiotic study, study 2, at baseline, change from the baseline at 12 weeks and change from baseline at 24 weeks.
Neuropsychology assessment: Memory Impairment Screen (MIS) | Baseline for all the group subjects subjects in microbiota composition study.
  Memory Impairment Screen (MIS). Screening test for memory impairment.
  At Baseline for no intervention study, study 1.
Neuropsychology assessment: Categorical Recall Test (Barcelona-2 Test) | Baseline for all the group subjects subjects in microbiota composition study.
  Categorical Recall Test (Barcelona-2 Test), semantic and phonemic fluency tests
  At Baseline for no intervention study, study 1.
Neuropsychology assessment: Orientation | Baseline for all the group subjects subjects in microbiota composition study.
  Orientation in Time, Space and Person (Barcelona-2 Test)
  At Baseline for no intervention study, study 1.
Neuropsychology assessment: Free and Cue Selective Reminding Test (FCSRT) | Baseline for all the group subjects subjects in microbiota composition study.
  Free and Cue Selective Reminding Test (FCSRT). Long and short Memory assessment test.
  At Baseline for no intervention study, study 1.
Neuropsychology assessment: Trial Making Test (TMT) A and B | Baseline for all the group subjects subjects in microbiota composition study.
  TMT A and B. Measures visuospatial, attention and executive functions.
  At Baseline for no intervention study, study 1.
Neuropsychology assessment: Boston Abbreviated Naming Test | Baseline for all the group subjects subjects in microbiota composition study.
  Boston Abbreviated Naming Test
  At Baseline for no intervention study, study 1.
Neuropsychology assessment: Verbal span | Baseline for all the group subjects subjects in microbiota composition study.
  Verbal Span (Barcelona-2 Test), that assesses attentional span and control/working memory.
  At Baseline for no intervention study, study 1.
Neuropsychology assessment: Clock test | Baseline for all the group subjects subjects in microbiota composition study.
  Clock Test, screening test for detecting cognitive impairment
  At Baseline for no intervention study, study 1.
Neuropsychology assessment: Frontal Assessment Battery (FAB) | Baseline for all the group subjects subjects in microbiota composition study.
  Frontal Assessment Battery (FAB), that assesses impairments related to frontal lobe function.
  At Baseline for no intervention study, study 1.
Neuropsychology assessment: Simple and semi complex constructive praxis (Barcelona-2 Test) | Baseline for all the group subjects subjects in microbiota composition study.
  Simple and semi complex constructive praxis (Barcelona-2 Test)
  At Baseline for no intervention study, study 1.
Neuropsychology assessment: Abbreviated Barcelona-2 Test | Baseline, change from baseline at 12 weeks and change from baseline at 24 weeks for AD patients in the probiotic study.
  Abbreviated Barcelona-2 Test. Abbreviated neuropsychological battery already normalised in Spanish populations.
  Only for the probiotic study, study 2, at baseline, change from baseline at 12 weeks and change from baseline at 24 weeks.
Neuropsychiatric assessment: Golberg Anxiety and Depression Scale | Baseline for all the group subjects subjects in microbiota composition study. Baseline, change from baseline at 12 weeks and change from baseline at 24 weeks for AD patients in the probiotic study.
  Golberg Anxiety and Depression Scale (more punctuation, more anxiety or depression symptoms) At Baseline for no intervention study
  For the probiotic study:
  At baseline, change from baseline at 12 weeks and change from baseline at 24 weeks.
Neuropsychiatric assessment: Neuropsychiatric Symptoms (Barcelona-2 Test) | Baseline for all the group subjects subjects in microbiota composition study. Baseline, change from baseline at 12 weeks and change from baseline at 24 weeks for AD patients in the probiotic study.
  For microbiota composition study, the following tests will be assessed:
  Neuropsychiatric Symptoms (Barcelona-2 Test), (more punctuation, more neuropsychiatric symptoms) At Baseline for no intervention study
  For the probiotic study:
  At baseline, change from baseline at 12 weeks and change from baseline 24 weeks.
Functional assessment | Baseline for all the group subjects subjects in microbiota composition study. Baseline, change from baseline at 12 weeks and change from baseline at 24 weeks for AD patients in the probiotic study.
  For microbiota composition study, the following tests will be assessed:
  Activities of Daily Living (ADL) (Barcelona-2 Test), (more punctuation, more dependent; punctuation total scale 0-100, Instrumental activities 0-60 + Basic activities 0-40) At Baseline for no intervention study
  For the probiotic study:
  At baseline, change from baseline at 12 weeks and change from baseline at 24 weeks, the following tests will be assessed:
  Activities of Daily Living ADL (Barcelona-2 Test), (more punctuation, more dependent; punctuation total scale 0-100, Instrumental activities 0-60 + Basic activities 0-40)

SECONDARY OUTCOMES:
Assessment of stress events | Baseline for all the group subjects subjects in microbiota composition study. Baseline, change from baseline at 12 weeks and change from baseline at 24 weeks for AD patients in the probiotic study.
  For microbiota composition study, the following tests will be assessed:
  Life Events Questionnaire, adapted from the Predimed-Plus study, which provides information on successfully overcome stressful events that could affect and modify the main variables under study (more punctuation, more stress).
  At Baseline for no intervention study
  For the probiotic study:
  At baseline, change from baseline at 12 weeks and change from baseline at24 weeks, the following tests will be assessed:
  Life Events Questionnaire, adapted from the Predimed-Plus study, which provides information on successfully overcome stressful events that could affect and modify the main variables under study (more punctuation, more stress).
Mediterranean lifestyle assessment | Baseline for all the group subjects subjects in microbiota composition study. Baseline, change from baseline at 12 weeks and change from baseline at 24 weeks for AD patients in the probiotic study.
  For microbiota composition study, the following tests will be assessed:
  Mediterranean lifestyle index interview (MEDLIFE), which provides information on how the patient follows the Mediterranean diet and lifestyle habits, more punctuation, more adhered to Mediterranean lifestyle.
  At Baseline for no intervention study
  For the probiotic study:
  At baseline, change from baseline at 12 weeks and change from baseline at24 weeks, the following tests will be assessed:
  Mediterranean lifestyle index interview (MEDLIFE), which provides information on how the patient follows the Mediterranean diet and lifestyle habits, more punctuation, more adhered to Mediterranean lifestyle.
Cognitive reserve assessment | Baseline for all the group subjects subjects in microbiota composition study. Baseline, change from baseline at 12 weeks and change from baseline at 24 weeks for AD patients in the probiotic study.
  For microbiota composition study, the following tests will be assessed:
  Cognitive reserve scale (more punctuation more cognitive reserve, score 0-25) At Baseline for no intervention study
  For the probiotic study:
  At baseline, change from baseline at 12 weeks and change from baseline at 24 weeks, the following tests will be assessed:
  Cognitive reserve scale (more punctuation more cognitive reserve, score 0-25)

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Torrente, Dr, Principal Investigator — University Rovira i Virgili
Locations (1):
- Dr. Margarita Torrente, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
It is not decided yet.

REFERENCES:
- [Background] Cabrera C, Vicens P, Torrente M. Modifiable Risk Factors for Dementia: The Role of Gut Microbiota. Curr Alzheimer Res. 2021;18(13):993-1009. doi: 10.2174/1567205018666211215152411. PMID 34911422
- [Background] Agahi A, Hamidi GA, Daneshvar R, Hamdieh M, Soheili M, Alinaghipour A, Esmaeili Taba SM, Salami M. Does Severity of Alzheimer's Disease Contribute to Its Responsiveness to Modifying Gut Microbiota? A Double Blind Clinical Trial. Front Neurol. 2018 Aug 15;9:662. doi: 10.3389/fneur.2018.00662. eCollection 2018. PMID 30158897
- [Background] Akbari E, Asemi Z, Daneshvar Kakhaki R, Bahmani F, Kouchaki E, Tamtaji OR, Hamidi GA, Salami M. Effect of Probiotic Supplementation on Cognitive Function and Metabolic Status in Alzheimer's Disease: A Randomized, Double-Blind and Controlled Trial. Front Aging Neurosci. 2016 Nov 10;8:256. doi: 10.3389/fnagi.2016.00256. eCollection 2016. PMID 27891089
- [Background] Benton D, Williams C, Brown A. Impact of consuming a milk drink containing a probiotic on mood and cognition. Eur J Clin Nutr. 2007 Mar;61(3):355-61. doi: 10.1038/sj.ejcn.1602546. Epub 2006 Dec 6. PMID 17151594
- [Background] Davari S, Talaei SA, Alaei H, Salami M. Probiotics treatment improves diabetes-induced impairment of synaptic activity and cognitive function: behavioral and electrophysiological proofs for microbiome-gut-brain axis. Neuroscience. 2013 Jun 14;240:287-96. doi: 10.1016/j.neuroscience.2013.02.055. Epub 2013 Mar 7. PMID 23500100
- [Background] Kelly JR, Allen AP, Temko A, Hutch W, Kennedy PJ, Farid N, Murphy E, Boylan G, Bienenstock J, Cryan JF, Clarke G, Dinan TG. Lost in translation? The potential psychobiotic Lactobacillus rhamnosus (JB-1) fails to modulate stress or cognitive performance in healthy male subjects. Brain Behav Immun. 2017 Mar;61:50-59. doi: 10.1016/j.bbi.2016.11.018. Epub 2016 Nov 16. PMID 27865949
- [Background] Messaoudi M, Lalonde R, Violle N, Javelot H, Desor D, Nejdi A, Bisson JF, Rougeot C, Pichelin M, Cazaubiel M, Cazaubiel JM. Assessment of psychotropic-like properties of a probiotic formulation (Lactobacillus helveticus R0052 and Bifidobacterium longum R0175) in rats and human subjects. Br J Nutr. 2011 Mar;105(5):755-64. doi: 10.1017/S0007114510004319. Epub 2010 Oct 26. PMID 20974015
- [Background] Saji N, Niida S, Murotani K, Hisada T, Tsuduki T, Sugimoto T, Kimura A, Toba K, Sakurai T. Analysis of the relationship between the gut microbiome and dementia: a cross-sectional study conducted in Japan. Sci Rep. 2019 Jan 30;9(1):1008. doi: 10.1038/s41598-018-38218-7. PMID 30700769
- [Background] Tillisch K, Labus J, Kilpatrick L, Jiang Z, Stains J, Ebrat B, Guyonnet D, Legrain-Raspaud S, Trotin B, Naliboff B, Mayer EA. Consumption of fermented milk product with probiotic modulates brain activity. Gastroenterology. 2013 Jun;144(7):1394-401, 1401.e1-4. doi: 10.1053/j.gastro.2013.02.043. Epub 2013 Mar 6. PMID 23474283
- [Background] Vogt NM, Kerby RL, Dill-McFarland KA, Harding SJ, Merluzzi AP, Johnson SC, Carlsson CM, Asthana S, Zetterberg H, Blennow K, Bendlin BB, Rey FE. Gut microbiome alterations in Alzheimer's disease. Sci Rep. 2017 Oct 19;7(1):13537. doi: 10.1038/s41598-017-13601-y. PMID 29051531
- [Background] Soldevila-Domenech N, Forcano L, Vintro-Alcaraz C, Cuenca-Royo A, Pinto X, Jimenez-Murcia S, Garcia-Gavilan JF, Nishi SK, Babio N, Gomis-Gonzalez M, Corella D, Sorli JV, Fernandez-Carrion R, Martinez-Gonzalez MA, Marti A, Salas-Salvado J, Castaner O, Fernandez-Aranda F, Torre R. Interplay between cognition and weight reduction in individuals following a Mediterranean Diet: Three-year follow-up of the PREDIMED-Plus trial. Clin Nutr. 2021 Sep;40(9):5221-5237. doi: 10.1016/j.clnu.2021.07.020. Epub 2021 Aug 5. PMID 34474192
- [Background] Buschke H. Cued recall in amnesia. J Clin Neuropsychol. 1984 Nov;6(4):433-40. doi: 10.1080/01688638408401233. PMID 6501581
- [Background] Buschke H, Kuslansky G, Katz M, Stewart WF, Sliwinski MJ, Eckholdt HM, Lipton RB. Screening for dementia with the memory impairment screen. Neurology. 1999 Jan 15;52(2):231-8. doi: 10.1212/wnl.52.2.231. PMID 9932936
- [Background] Dubois B, Slachevsky A, Litvan I, Pillon B. The FAB: a Frontal Assessment Battery at bedside. Neurology. 2000 Dec 12;55(11):1621-6. doi: 10.1212/wnl.55.11.1621. PMID 11113214
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Goldberg D, Bridges K, Duncan-Jones P, Grayson D. Detecting anxiety and depression in general medical settings. BMJ. 1988 Oct 8;297(6653):897-9. doi: 10.1136/bmj.297.6653.897. PMID 3140969
- [Background] Hughes CP, Berg L, Danziger WL, Coben LA, Martin RL. A new clinical scale for the staging of dementia. Br J Psychiatry. 1982 Jun;140:566-72. doi: 10.1192/bjp.140.6.566. PMID 7104545
- [Background] Pena-Casanova J, Quinones-Ubeda S, Gramunt-Fombuena N, Aguilar M, Casas L, Molinuevo JL, Robles A, Rodriguez D, Barquero MS, Antunez C, Martinez-Parra C, Frank-Garcia A, Fernandez M, Molano A, Alfonso V, Sol JM, Blesa R; NEURONORMA Study Team. Spanish Multicenter Normative Studies (NEURONORMA Project): norms for Boston naming test and token test. Arch Clin Neuropsychol. 2009 Jun;24(4):343-54. doi: 10.1093/arclin/acp039. Epub 2009 Aug 1. PMID 19648582
- [Background] Reisberg B. Functional assessment staging (FAST). Psychopharmacol Bull. 1988;24(4):653-9. No abstract available. PMID 3249767
- [Background] Reisberg B, Ferris SH, de Leon MJ, Crook T. The Global Deterioration Scale for assessment of primary degenerative dementia. Am J Psychiatry. 1982 Sep;139(9):1136-9. doi: 10.1176/ajp.139.9.1136. PMID 7114305
- [Background] REITAN RM. The relation of the trail making test to organic brain damage. J Consult Psychol. 1955 Oct;19(5):393-4. doi: 10.1037/h0044509. No abstract available. PMID 13263471
- [Background] Shulman KI. Clock-drawing: is it the ideal cognitive screening test? Int J Geriatr Psychiatry. 2000 Jun;15(6):548-61. doi: 10.1002/1099-1166(200006)15:63.0.co;2-u. PMID 10861923
- [Background] Sotos-Prieto M, Santos-Beneit G, Bodega P, Pocock S, Mattei J, Penalvo JL. VALIDATION OF A QUESTIONNAIRE TO MEASURE OVERALL MEDITERRANEAN LIFESTYLE HABITS FOR RESEARCH APPLICATION: THE MEDITERRANEAN LIFESTYLE INDEX (MEDLIFE). Nutr Hosp. 2015 Sep 1;32(3):1153-63. doi: 10.3305/nh.2015.32.3.9387. PMID 26319833
- See also: Pena-Casanova J. (2019). Teoria e Interpretacion: Normalidad, Semiologia y Patologia Neuropsicologicas. Programa integrado de exploracion neuropsicologica. Test Barcelona-2. Masquelibros, S.L., Jaen. International Standrad Book Number: 978-84-120274-0-2. — https://www.test-barcelona.com/es/

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/25/NCT05943925/Prot_SAP_000.pdf
  • Informed Consent Form: study 1 (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT05943925/ICF_001.pdf
  • Informed Consent Form: study 2 (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT05943925/ICF_002.pdf